CLINICAL TRIAL: NCT02866812
Title: Prevalence and Factors Associated With the Occurrence of Depression Six Months After an Endovascular Treatment of Intracranial Aneurysm
Acronym: DEP-AIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PA15099
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

ARMS (1):
- patient with endovascular treatment for intracranial aneurysm (Experimental)
  Interventions: Other: questionnaires assessing the state of fatigue, depression and anxiety

INTERVENTIONS:
Other: questionnaires assessing the state of fatigue, depression and anxiety

SUMMARY:
During the last decade, the embolization has become the treatment of choice for ruptured intracranial aneurysms, to improve the neurological outcome of patients. At the same time, for his safety, she also became the technique allowing prophylactic treatment of unruptured intracranial aneurysms discovered incidentally during imaging exams.

Regarding patients with ruptured intracranial aneurysms, patients who survive often have a reduced quality of life while one in two has a good neurological outcome after embolization. Depression, anxiety and fatigue, whose the psycho-social impact is important, are often cited. This description has often been done without considering the realized type of treatment (surgery or embolization) and mostly of neurological and functional status of the patient remotely (disability or not in daily activities).

Regarding patients with unruptured intracranial aneurysms, they are mostly asymptomatic and embolization is programmed. They would present an cognitive impairment in one case in five at 1 month of treatment.

If depression, fatigue and difficult return to working life are logically found in patients with severe sequelae (disability in daily activities) of their ruptured intracranial aneurysms, the question arises for patients with a ruptured intracranial aneurysms with a favorable evolution and for asymptomatic patients with unruptured intracranial aneurysms.

A precise status of these populations is necessary, especially as the discovery and treatment of their intracranial aneurysms is often early (between 40 and 60 years) and that their good neurological status should allow "a priori" to return easily at the active life.

DETAILED DESCRIPTION:
Describe the prevalence of depression among patients treated for intracranial aneurysms, especially in patients with a favorable neurological outcome at 6 months (mRS inferior or egal to 1).

Study factors associated with the presence of depression in patients treated for intracranial aneurysms, especially in patients with a favorable neurological outcome at 6 months (mRS inferior or egal to 1)

ELIGIBILITY:
Inclusion Criteria:

* patient with endovascular treatment for intracranial aneurysm (ruptured or unruptured)
* patient older than 18 years
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program

Exclusion Criteria:

* patient with anterior treatment for intracranial aneurysm
* bipolar disorder, schizophrenia or schizoaffective disorder diagnostic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
depression | 6 months
  Depression evaluated using the Hamilton scale

SECONDARY OUTCOMES:
tired | 6 months
  tired evaluated using the Piper scale
anxiety | 6 months
  tired evaluated using the State - Trait Anxiety Inventory Form Y

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France